CLINICAL TRIAL: NCT02063971
Title: Tolerance and Efficacy Evaluation of Three Face Creams in Subjects Undergoing to Injection Procedure With Hyaluronic Acid (Intradermal Implant)
Brief Title: Tolerance and Efficacy Evaluation of 3 Face Creams
Acronym: FILLER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adele Sparavigna (Other)
Responsible Party: Sponsor-Investigator, Adele Sparavigna, Physician, Derming SRL
Organization: Derming SRL (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E3513 / SC13-235
Record Dates: First submitted 2014-02-07; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Skin Aging
Keywords: Skin aging; Soothing activity; Hyaluronic acid injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin aging (Experimental): Anti-age product will be applied once a day, in the evening, on half face and neck for an uninterrupted period of 12 weeks and the placebo cream in the morning with the same modalities. On the contralateral face side (right or left side according to a previous randomisation list), the volunteers will apply the placebo cream twice a day
  Interventions: Other: Soothing (formulation number: F#1048-082) and antiaging creams (F#841-020 and F#1374-002)

INTERVENTIONS:
Other: Soothing (formulation number: F#1048-082) and antiaging creams (F#841-020 and F#1374-002)

SUMMARY:
The study will evaluate the tolerance and the efficacy on skin comfort of F#1048-082 soothing cream used just after injection procedure and also the tolerance and the efficacy of the F#841-020 anti-age cream on aging parameters compared to baseline and to the F#1374-002 placebo cream (comparison within subjects - half face method) to identify additional benefits delivered by the product compared to a cosmetic procedure.

DETAILED DESCRIPTION:
First study phase (soothing activity)

* Clinical grading (visual analogic scale):

  1. Erythema (0= no erythema to 10= strong erythema)
  2. Oedema (0= no oedema to 10= strong oedema)
  3. Bruise (0= no bruise to 10= strong bruise)
  4. Overall skin appearance (0= bad overall appearance to 10= good overall appearance).
* Optical colorimetry: measurement of redness/bruise (L*a*b*) by Spectrophotometer CM-2600d.
* Photographic documentation: Canfield imaging station equipped with visible, polarized, fluorescence and UV light and with specific lighting for shadows.

Second study phase (anti-age activity vs placebo):

* Clinical and self grading (visual analogic scale) :

  1. Forehead wrinkles (0= no wrinkle to 10= severe wrinkles)
  2. Crow's feet wrinkles (0= no wrinkle to 10= severe wrinkles)
  3. Crow's feet fine lines (0= no fine line to 10= severe fine lines)
  4. Under the eye wrinkles (0= no wrinkle to 10= severe wrinkles)
  5. Under the eye fine lines (0= no fine line to 10= severe fine lines)
  6. Frown lines (0= no wrinkle to 10= severe wrinkles)
  7. Marionette lines (0= no wrinkle to 10= severe wrinkles)
  8. Upper lip wrinkles (0= no wrinkle to 10= severe wrinkles)
  9. Nasolabial folds (0= no wrinkle to 10= severe wrinkles)
  10. Cheek wrinkles (0= no wrinkle to 10= severe wrinkles)
  11. Neck wrinkles (0= no wrinkle to 10= severe wrinkles)
  12. Lines on the neck opening (0= no wrinkle to 10= severe wrinkles)
  13. Skin firmness (0= very firm skin to 10= no firm skin)
  14. Skin elasticity (0= very elastic skin to 10= no elastic skin)
  15. Sagging skin (0= no sagging skin to 10= severe sagging skin)
  16. Radiance (0= very radiant skin to 10= no radiant skin)
  17. Smoothness (0= very smooth skin to 10= no smooth skin)
  18. Skin softness (0= very soft skin to 10= no soft skin)
  19. Colour evenness (0= good evenness to 10= bad evenness)
  20. Skin tone (0= good complexion to 10= bad complexion)
* Optical colorimetry: measurement of skin colour (L*a*b*) by Spectrophotometer CM-2600d.
* Photographic documentation: Canfield imaging station equipped with visible, polarized, fluorescence and UV light and with specific lighting for shadows.
* Skin replicas and profilometry at level of crow's feet (image analysis of: total surface of the wrinkles, mean length of the wrinkles, total length of the wrinkles, number of the wrinkles)
* Skin elasticity measurement by suction (Cutometer®)

Tolerance evaluation (investigator's judgement):

At each evaluation time, the investigator considering the appearance of possible adverse effects related to the tested creams and all comments reported by the subjects on diary card will judge the tolerance of the products under study.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* age > 35 years old
* good general state of health
* woman who had already undergone Hyaluronic acid injections
* woman who have not applied any retinoid product in the last 3 months
* woman who are not in a recovery period after laser/peeling/acne treatment
* accepting to return to the centre for the planned visits
* accepting to follow the investigator's instructions during the entire study period
* agreeing to present at each study visit without make-up
* accepting to not change their habits regarding: food, physical activity, face cleansing and make-up use
* agreeing to not receive any drug able to change the skin characteristics during the entire duration of the study
* accepting to not receive any cutaneous anti-age treatment during the entire duration of the study
* accepting not to expose their face to strong UV irradiation (UV session or sun bathes) during the entire duration of the study
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Pregnancy (only for subjects not in menopause)
* lactation (only for subjects not in menopause)
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test during the basal visit (T0), 6 and 12 weeks after the intradermal implant execution;
* subjects participating to a similar test less than 3 months ago
* sensitivity to the test products or theirs ingredients
* subjects whose insufficient adhesion to the study protocol is foreseeable.
* dermatitis
* presence of cutaneous disease on the tested area as lesions, scars, malformations.
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.)
* recurrent facial/labial herpes.
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* digestive disease
* haematological disease
* chronic phlogosis or autoimmune disease
* cancer
* neurological or psychological disease
* drug allergy.
* systemic corticosteroids
* retinoid products in the previous 3 months and during the entire study period
* aspirin or non-steroid anti-inflammatory drugs (FANS)
* anti-histaminic, narcotic, antidepressant, immunosuppressive drugs (with except, for female subjects, of contraceptive or hormonal treatment starting from at least one year)
* assumption of drugs able to influence the test results in the investigator opinion.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Tolerance and the efficacy on skin comfort of F#1048-082 soothing cream used just after injection procedure on nasolabial folds | 1 week
  For 7 days after injections (from T0 to T7d/T0'') the soothing cream will be applied twice a day on the full face and neck insisting on injection areas. 5 visits will be performed: a pre-test visit (T-30 subjects' screening), a baseline visit (T0 intradermal implant execution/ T0' evaluations just after the aesthetic procedure/ Timm evaluations immediately after the 1st soothing cream application), 2 intermediate visits (T1d, T3d - 1 and 3 days after injections) and a final visit (T7d - 7 days after the aesthetic procedure). Product tolerance (number of participants with adverse events) and efficacy:
  * clinical and self grading (performed on injection areas by VAS score)
  * optical colorimetry (on nasolabial folds - L*a*b*)
  * photographic documentation (of all the face) will be performed at each study time.

SECONDARY OUTCOMES:
Evaluation of the tolerance and the efficacy of the F#841-020 anti-age cream on aging parameters compared to baseline and to the F#1374-002 placebo cream to identify additional benefits delivered by the product compared to a cosmetic procedure | 3 months
  The anti-age product will be applied once a day, in the evening, on half face and neck, for 12 weeks and the placebo cream in the morning with the same modalities. On the contralateral face side (according to a previous randomisation list), the volunteers will apply the placebo cream twice a day.
  5 visits will be performed: a baseline visit (T0 - before aesthetic procedure), a visit 7 days after injection (T0''/T7d), 2 intermediate visits (T4W and T8W - 4 and 8 weeks after the first study product application) and a final visit (T12W - 12 weeks after the first study product application).
  Tolerance (number of participants with adverse events) and efficacy:
  * clinical and self grading on face and neck (by VAS score)
  * optical colorimetry on both cheeks (L*a*b*)
  * photographic documentation of all the face
  * skin elasticity on both cheeks (deformation-mm)
  * wrinkles profilometry on the lateral corner of the eyes (micron) will be evaluated at each study time.

CONTACTS AND LOCATIONS:
Overall Officials: ADELE SPARAVIGNA, PHYSICIAN, Principal Investigator — Derming SRL
Locations (1):
- DERMING, Monza, Monza-brianza, Italy